CLINICAL TRIAL: NCT01305005
Title: To Investigate Ocular Haemodynamics After Phacoemulsification Surgery
Brief Title: Effect of Phacoemulsification on Ocular Blood Flow in Human
Status: Completed | Type: Observational
Sponsor: yin ying zhao (Other)
Responsible Party: Sponsor-Investigator, yin ying zhao, Yin Ying Zhao, Wenzhou Medical University
Organization: Wenzhou Medical University (Other)
Other Study IDs: WZMC2011BNZYJ
Record Dates: First submitted 2011-02-25; First posted 2011-02-28 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Cataract; Hypertension; Diabetes
Keywords: blood flow
MeSH Terms: conditions — Cataract; Hypertension; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients with active-fluidics system: patients who underwent phacoemulsification surgery using active-fluidics system
- patients with gravity-fluidics system.: patients who underwent phacoemulsification surgery using gravity-fluidics system

SUMMARY:
* To investigate ocular haemodynamics after phacoemulsification surgery
* To evaluate the influence in people with different autoregulation of ocular blood flow

ELIGIBILITY:
Inclusion Criteria:

* age-related cataract
* no complications during surgery

Exclusion Criteria:

* complications during surgery
* have other complications

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients who underwent phacoemulsification surgery in Eye Hospital of Wenzhou Medical College
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2011-03; Primary Completion 2018-11 (Actual); Study Completion 2019-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: qu jia, MD, Principal Investigator — Wenzhou Medical University
Locations (1):
- Eye Hospital of Wenzhou Medical College, Wenzhou, Zhejiang, China

REFERENCES:
- [Derived] Zhao Y, Wang D, Nie L, Yu Y, Zou R, Li Z, Xu M, Zhao Y. Early changes in retinal microcirculation after uncomplicated cataract surgery using an active-fluidics system. Int Ophthalmol. 2021 May;41(5):1605-1612. doi: 10.1007/s10792-021-01694-4. Epub 2021 Feb 6. PMID 33547997